CLINICAL TRIAL: NCT01631266
Title: A Phase III Contact Tracing Trial Comparing the Diagnostic Performance of C-Tb to QuantiFERON®-TB Gold In-Tube, in Combination With a Double Blind Randomized Split Body Safety Assessment of C-Tb Versus 2 T.U. Tuberculin PPD RT23 SSI
Brief Title: Comparison of Diagnostic Performance of C-Tb to QuantiFERON®-TB, in Combination With a Safety Assessment of C-Tb vs Tuberculin PPD RT23 SSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: TESEC-06; 2011-005617-36 (EudraCT Number)
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.1 µg/0.1 mL C-Tb (Experimental): The C-Tb and 2 T.U. Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT and LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: C-Tb
- 2 T.U. Tuberculin PPD RT 23 SSI (Active Comparator): The C-Tb and 2 T.U. Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT and LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: 2 T.U. Tuberculin PPD RT 23 SSI

INTERVENTIONS:
Biological: C-Tb — The C-Tb agent is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearm according to a double blind randomisation scheme
  Arms: 0.1 µg/0.1 mL C-Tb
Biological: 2 T.U. Tuberculin PPD RT 23 SSI — The 2 T.U. Tuberculin PPD RT 23 SSI agent is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearm according to a double blind randomisation scheme
  Arms: 2 T.U. Tuberculin PPD RT 23 SSI

SUMMARY:
Tuberculosis (TB) continues to be the most important bacterial infection worldwide and therefore new improved diagnostic tests are needed to help doctors in diagnosing TB.

We are investigating a new skin test named C-Tb. Like the current tuberculin skin test (PPD), the C-Tb test is injected just under the skin and will, when positive, show redness and/or swelling at the injection site while a negative test will leave no reactions.

The aim of this trial is to test the C-Tb skin test in volunteers. The volunteers are divided into four groups:

* Negative control group: Must have no history of exposure to a person with tuberculosis disease.
* Occasional contact: Must be in contact with a person with tuberculosis disease between 6 hours/week and 6 hours/day
* Close contact: Must be in close contact with a person with tuberculosis disease for more than 6 hours/day for at least five days
* Positive control group: Must have a confirmed tuberculosis disease within the last 3 years.

The goals of this clinical trial are:

* To compare the C-Tb test to a blood test, the QuantiFERON test.
* To compare the C-Tb test to the PPD test that is currently being used.
* To assess the safety of the C-Tb test.

DETAILED DESCRIPTION:
The TESEC-06 trial is an open comparison of the diagnostics performance of C-Tb compared to QuantiFERON®-TB Gold In-Tube, in combination with a double-blind randomized split-body safety assessment of C-Tb versus Tuberculin PPD RT23 SSI.

The trial is designed to address the fundamental issue that in the diagnosis of latent tuberculosis (TB) infection, no gold standard exists. Thus, no existing test for latent TB is 100 % sensitive and specific - including the Tuberculin PPD RT23 SSI and QuantiFERON®-TB Gold In-Tube.

This will be addressed by evaluating C-Tb positive response rates in 4 groups defined by their estimated risk of infection with MTb. The groups will consist of paediatric and adult participants selected as being either occasional or close contacts to an active pulmonary TB case. In addition a group of confirmed TB cases and a group of participants with no history of exposure to MTb will be included as control groups.

50 participants in the negative control group will be tested with C-Tb alone in order to evaluate whether concomitant administration of C-Tb and Tuberculin PPD RT23 SSI could conceivably result in larger or smaller areas of induration to one or both tests as a result of expanding the clone of sensitised T-cells i.e. since Tuberculin PPD RT23 SSI includes among several other antigens ESAT-6 and CFP-10 and C-Tb also contains both these antigens.

ELIGIBILITY:
Inclusion Criteria:

1. Can comply with one of the following groups:

   1. Negative control group: Must have no history of exposure to a TB index case, and have no signs or symptoms of TB
   2. Positive control group: Confirmed TB disease within the last 3 years by sputum smear microscopy and/or Culture, Gene Xpert or PCR
   3. Close contact group: Must be in close contact with a pulmonary smear positive TB index case for more than 6 hours/day for at least five days
   4. Occasional contact group: Must be in contact with a pulmonary sputum smear positive TB index case between 6 hours/week and 6 hours/day
2. Is between 6 weeks - 65 years of age
3. Participant, parent or legal guardian has provided signed informed consent
4. Is willing and likely to comply with the trial procedures
5. Is prepared to grant authorized persons access to their medical records

Exclusion Criteria:

1. Has been vaccinated with a live vaccine within 6 weeks prior to the day of inclusion (e.g. Mumps Measles Rubella (MMR), yellow fever, oral typhoid vaccines)
2. Has been tuberculin tested less than 12 months prior to the day of inclusion
3. Is pregnant, breastfeeding or intending to get pregnant within the trial period
4. Is a female of child bearing potential (12 years of age or older having had their first menstruation) not willing to use effective barrier (including spermicidal gel), hormonal or intrauterine contraceptive measures within the trial period
5. Has an active disease affecting the lymphoid organs except for HIV (e.g., Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
6. Has a current skin condition which interferes with the reading of the C-Tb and Tuberculin PPD RT23 SSI e.g. tattoos, severe scarring, burns/sunburns, rash, eczema, psoriasis, or any other skin disease at or near the injection sites
7. Has a condition where blood drawings pose more than minimal risk for the participant, such as haemophilia, other coagulation disorders, or significantly impaired venous access
8. Current participation in another clinical trial with an investigational or non investigational drug or device, which in the opinion of investigator may interfere with this trial drug
9. Has participated in previous clinical trials investigating injections with ESAT-6 and/or CFP-10 antigens
10. Has a condition which in the opinion of the investigator is not suitable for participation in the trial

Ages: 6 Weeks to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate an increasing trend in C-Tb test positivity across the four study groups, with 'positivity' defined as an induration ≥ 5 mm | Onset between the injections and 28 days after the injections

SECONDARY OUTCOMES:
To demonstrate a significantly lower response rate of C-Tb as compared to that of PPD RT23 SSI in the BCG vaccinated participants in the negative control group, with response defined as any induration (> 1mm) for both agents | Onset between the injections and 28 days after the injections
To evaluate a possible trend in C-Tb induration diameters across the four pre-specified MTb infection risk sub-groups | Onset between the injections and 28 days after the injections
To evaluate a possible trend in PPD RT23 SSI induration diameters across the four pre-specified MTb infection risk sub-groups | Onset between the injections and 28 days after the injections
To evaluate a possible trend in QuantiFERON Gold In-Tube results across four pre-specified MTb infection risk sub-groups | On the day of the injections
To evaluate a possible trend in PPD RT23 SSI test positivity across four pre-specified MTb infection risk sub-groups | Onset between the injections and 28 days after the injections
To evaluate a possible trend in QuantiFERON Gold In-Tube test positivity across four pre-specified MTb infection risk sub-groups | On the day of the injections
To evaluate the difference in sensitivity between C-Tb and QuantiFERON Gold In-Tube in the positive control group | From the day of injections to 2-3 days after the injections
To evaluate the difference in specificity between C-Tb and QuantiFERON Gold In-Tube in the negative control group | From the day of injections to 2-3 days after the injections
To evaluate the difference in sensitivity between C-Tb and PPD RT23 SSI in positive control group | Onset between the injections and 28 days after the injections
To evaluate the difference in specificity between C-Tb and PPD RT23 SSI in the negative control group | Onset between the injections and 28 days after the injections
To compare the size of induration of C-Tb if injected alone or concomitantly with PPD RT23 SSI in negative control group | Onset between the injections and 28 days after the injections
To compare the specificity of C-Tb if injected alone or concomitantly with PPD RT23 SSI, in the negative control group | Onset between the injections and 28 days after the injections
To compare the diagnostic outcome of C-Tb to that of QuantiFERON Gold In-Tube using a latent class approach | From the day of injections to 2-3 days after the injections
To compare the diagnostic outcome of C-Tb to that of PPD RT23 SSI using a latent class approach | Onset between the injections and 28 days after the injections
To evaluate the secondary analyses above (1-14) of C-Tb and PPD RT23 SSI using alternative cut-off values | Onset between the injections and 28 days after the injections
To compare the diagnostic outcome of C-Tb and QuantiFERON Gold In-Tube stratified on the four study groups | From the day of injections to 2-3 days after the injections
To compare the diagnostic outcome of C-Tb and PPD RT23 SSI stratified on the four study groups | Onset between the injections and 28 days after the injections
To evaluate the clinical safety of C-Tb | Onset between the injections and 28 days after the injections
To evaluate the clinical safety of PPD RT23 SSI | Onset between the injections and 28 days after the injections

CONTACTS AND LOCATIONS:
Overall Officials: Joan Cayla, MD, Principal Investigator — Public Health Agency of Barcelona; Henrik Aggerbeck, M. Sc., Study Chair — Statens Serum Institut
Locations (13):
- Spain (13):
  - Hospital Universitario de Cruces, Barakaldo, Basque Country
  - CAP Drassanes, Unitat de Prevenció i Control de Tuberculosi, Barcelona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Public Health Agency of Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital Clínic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Mutua de Terrassa, Barcelona, Catalonia
  - Hospital San Joan De Deu, Barcelona, Catalonia
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Complexo Hospitalario de Pontevedra, Pontevedra, Galicia
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, Galicia
  - Complexo Hospitalario Universitario de Vigo, Vigo, Galicia

REFERENCES:
- [Derived] Ruhwald M, Aggerbeck H, Gallardo RV, Hoff ST, Villate JI, Borregaard B, Martinez JA, Kromann I, Penas A, Anibarro LL, de Souza-Galvao ML, Sanchez F, Rodrigo-Pendas JA, Noguera-Julian A, Martinez-Lacasa X, Tunez MV, Fernandez VL, Millet JP, Moreno A, Cobos N, Miro JM, Roldan L, Orcau A, Andersen P, Cayla JA; TESEC Working Group. Safety and efficacy of the C-Tb skin test to diagnose Mycobacterium tuberculosis infection, compared with an interferon gamma release assay and the tuberculin skin test: a phase 3, double-blind, randomised, controlled trial. Lancet Respir Med. 2017 Apr;5(4):259-268. doi: 10.1016/S2213-2600(16)30436-2. Epub 2017 Feb 1. PMID 28159608